CLINICAL TRIAL: NCT02063802
Title: Effect of an Intervention Program With Healthy Habits Plus Metformin or Conjugated Linoleic Acid Over Clinical Parameters and Molecular Pathways of Insulin Resistance in Obese Pediatric Patients
Brief Title: Metformin vs Conjugated Linoleic Acid and an Intervention Program With Healthy Habits in Obese Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Collaborators: Hospital General de Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DI/11/311/04/108
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
Keywords: pediatric obesity; conjugated linoleic acid; CLA; metformin
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Metformin; Linoleic Acids, Conjugated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- metformin and healthy habits program (Active Comparator): 1 gr per day. (250mg tablets). The patient takes 2 tablets with breakfast and 2 tablets with dinner and 2 placebo tablets with food by mouth for four months.
  Interventions: Drug: metformin; Behavioral: Healthy habits program
- Conjugated Linoleic Acid and healthy habits (Experimental): Total dose: 3gr per day (500mg capsules). The patient takes 2 capsules with breakfast, 2 capsules with lunch and 2 capsules with dinner by mouth for four months.
  Interventions: Dietary Supplement: Conjugated Linoleic Acid; Behavioral: Healthy habits program
- Placebo and healthy habits program (Placebo Comparator): Total dose 6 tablets per day. The patient takes 2 tablets with breakfast, two tablets with lunch and two tablets with dinner by mouth for four months.
  Interventions: Drug: Placebo; Behavioral: Healthy habits program

INTERVENTIONS:
Drug: metformin — total dose: 1 gr per day (250mg tablets). The patient takes 2 tablets with breakfast and 2 tablets with dinner and 2 placebo tablets with food by mouth for four months.
  Arms: metformin and healthy habits program
Dietary Supplement: Conjugated Linoleic Acid — total dose: 3gr/día(500mg capsules). The patient takes 2 capsules with breakfast, 2 capsules with lunch and 2 capsules with dinner for four months.
  Arms: Conjugated Linoleic Acid and healthy habits
Drug: Placebo — Total dose 6 tablets per day. The patient takes 2 tablets with breakfast, two tablets with lunch and two tablets with dinner by mouth for four months
  Arms: Placebo and healthy habits program
Behavioral: Healthy habits program

SUMMARY:
The purpose of this clinical trial is to examine the effects of conjugated linoleic acid (CLA) vs metformin along with an intervention program with healthy habits on body composition, weight, M value in CLAMP and clinical laboratory values, as well as molecular and genetic changes in obese children.

Patients from the pediatric service of the Hospital from 8 to 18 years old with a body mass index ≥ Pc 95 and 35kg/m2 are randomized to either interventional group for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between 8 and 18 years old
* Pc BMI ≥ 95 and <35kg/m2,
* No endocrine diseases, including diabetes mellitus
* No systemic diseases
* No genetic diseases
* No pharmacological treatment affecting lipid metabolism or glucose
* No history of acute or prolonged immobilization
* Normal aminotransferases
* Signed Informed consent and assent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body mass index at 4 months | baseline, 4 months
Change in body fat mass at 4 months | baseline, 4 months
Change in lean body mass at 4 months | baseline, 4 months

SECONDARY OUTCOMES:
Change in clinical laboratory values at 4 months | baseline, 4 months
Change in M Value in CLAMP at 4 months | baseline, 4 months
Change in muscle tissue transcriptome at 4 months | baseline, 4 months
Change in adipose tissue transcriptome at 4 months | baseline, 4 months
Change in inflammatory cytokines al 4 months | baseline, 4 months
Change in the phosphorylation of the insulin receptor in muscle tissue at 4 months | baseline, 4 months
Change in the phosphorylation of the insulin receptor in adipocytes at 4 months | baseline, 4 months
Change in activation status of proteins involved in insulin signaling of myocytes cDNA at 4 months | baseline, 4 months
Number of Participants with Serious and Non-Serious Adverse Events | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nayely G Garibay, Pediatrician, Principal Investigator — Hospital General de México; Gloria E Queipo, M.Specialist, Principal Investigator — Hospital General de México
Locations (1):
- General Hospital of Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Garibay-Nieto N, Queipo-Garcia G, Alvarez F, Bustos M, Villanueva E, Ramirez F, Leon M, Laresgoiti-Servitje E, Duggirala R, Macias T, Cuevas S, Jalife A, Fonseca-Sanchez M, Serratos F, Lopez-Alvarenga JC. Effects of Conjugated Linoleic Acid and Metformin on Insulin Sensitivity in Obese Children: Randomized Clinical Trial. J Clin Endocrinol Metab. 2017 Jan 1;102(1):132-140. doi: 10.1210/jc.2016-2701. PMID 27778642